CLINICAL TRIAL: NCT03142152
Title: Assessment of the Carillon Mitral Contour System® in Treating Heart Failure With at Least Mild Functional Mitral Regurgitation
Brief Title: The EMPOWER Trial - The Carillon Mitral Contour System® in Treating Heart Failure With at Least Mild FMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiac Dimensions, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cardiac Dimensions Pty Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVP 1670-01
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Functional Mitral Regurgitation; Heart Failure; Mitral Valve Insufficiency; Heart Diseases; Cardiovascular Diseases; Heart Valve Diseases
Keywords: Functional Mitral Regurgitation; Percutaneous Mitral Valve Repair; Percutaneous Mitral Valve Annuloplasty; Coronary Sinus Annuloplasty; Secondary Mitral Regurgitation; Functional MR; FMR
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency; Heart Diseases; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention Group (Experimental): Carillon Mitral Contour System and Guideline Directed Heart Failure Medication
  Interventions: Device: Carillon Mitral Contour System; Other: Guideline Directed Heart Failure Medication
- Control Group (Active Comparator): Guideline Directed Heart Failure Medication
  Interventions: Other: Guideline Directed Heart Failure Medication

INTERVENTIONS:
Device: Carillon Mitral Contour System — The Carillon implant is designed to be deployed, tensioned, and locked in the coronary vein in order to reshape the mitral annulus and thus reduce mitral annular dilation and mitral regurgitation.
  Other Names: Carillon; Percutaneous mitral valve repair
  Arms: Intervention Group
Other: Guideline Directed Heart Failure Medication — Heart failure medication per ACC/AHA guidelines

SUMMARY:
The objective of this prospective, randomized, blinded clinical trial is to assess the safety and efficacy of the Carillon Mitral Contour System in treating heart failure with functional regurgitation (FMR).

DETAILED DESCRIPTION:
A total of 300 subjects will be randomized at up to 75 investigational sites in the United States, Canada, and Europe. Subjects will be randomized into one of two study groups using a 1:1 (Intervention : Control) ratio.

Study subjects who are eligible for this clinical study will undergo a transthoracic echocardiographic examination prior to randomization to evaluate the inclusion criteria associated with the severity of mitral regurgitation. A coronary angiogram will be performed to evaluate the coronary artery anatomy and a venogram to assess the suitability of the coronary sinus/great cardiac vein (CS/GCV) for placement of the Carillon implant.

If the subject meets the anatomic requirements for device placement, the subject will be randomized. Subjects who meet all eligibility criteria will be randomized into one of two study groups (Intervention or Control).

Subjects randomized to the Intervention group will undergo the Carillon implant procedure.

Subjects randomized to the Control group will experience an index procedure similar to the Intervention group (without device placement) to ensure they will not be able to deduce the group assignment based on the type of intervention or time associated with the procedure.

After the study subjects are discharged, the subjects' primary care specialists (cardiologist/heart failure physician) and clinical investigation site staff will coordinate follow-up evaluations. Subjects will be evaluated at one (1), six (6), twelve (12), eighteen (18) and twenty-four (24) months post-randomization, to assess long-term safety, and functional and clinical status.

After the 24-month evaluation, all subjects will be unblinded. All Intervention and Control subjects will be followed with an abbreviated annual contact and echocardiogram for an additional three (3) years, for a total of five (5) years.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic heart failure with functional (secondary) mitral regurgitation of at least 1+ (mild) severity
2. NYHA II, III, or IV
3. Six Minute Walk distance ≥ 100 meters and ≤ 600 meters
4. Left Ventricular Ejection Fraction ≤ 50%
5. LVEDD ≥ 57 mm and LVESD ≤ 75 mm
6. Corrected BNP of > 300 pg/ml, or corrected NT-proBNP > 1200 pg/ml, or one or more heart failure hospitalizations within one year prior to consent
7. Guideline directed heart failure medication regimen
8. Age 18 years old
9. Carillon implant can be sized and placed in accordance with the IFU
10. The subject has been informed of the nature of the trial and agrees to its provisions, including the possibility of randomization to the Control group and returning for all required post-procedure follow-up visits, and has provided written informed consent

Exclusion Criteria:

1. Pre-existing device (e.g., pacing lead) in coronary sinus (CS) / great cardiac vein (GCV) or Class I indication for cardiac resynchronization therapy (CRT)
2. Presence of a mechanical or bio-prosthetic mitral valve or, mitral valve annuloplasty, or leaflet repair device
3. Significant organic mitral valve pathology (e.g., moderate or severe myxomatous degeneration, with or without mitral leaflet prolapse, rheumatic disease, full or partial chordal rupture)
4. Severe tricuspid regurgitation associated with right ventricular dysfunction and enlargement
5. Severe mitral annular calcification
6. Severe aortic stenosis
7. Expected to require any cardiac surgery, including surgery for coronary artery disease (CAD) or valve disease within one (1) year
8. Chronic, severe, medical conditions or pathology, other than heart failure, that will prevent likely survival beyond twelve (12) months or any other medical condition that, in the judgment of the Investigator, makes the patient a poor candidate for this study

   * An entire list of eligibility is available in the clinical investigational plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Objective - Freedom from Major Adverse Events | 12 months
  Freedom from a composite of major adverse events (defined as Device Embolization, Vessel Erosion, Cardiac Perforation, and occurrence of cardiac surgery or percutaneous coronary intervention) in the Intervention group is greater than performance goal of 90%.
Primary Efficacy Objective 1 - Hierarchical Clinical Composite | 24 months
  To demonstrate that the Carillon Mitral Contour System (Intervention) group is superior to the Control group on the hierarchical composite endpoint of death, transplant or LVAD, percutaneous or surgical mitral valve intervention, heart failure hospitalization, Improvement in KCCQ, and improvement in six-minute walk distance at 24 months (analyzed when the last subject completes 12 months of follow-up.)

SECONDARY OUTCOMES:
Secondary Efficacy Objective 1- Regurgitant Volume | 12 months
  To compare regurgitant volume change relative to control from baseline through 12 months of follow up
Secondary Efficacy Objective 2 - Change in LV End-diastolic Volume | 12 months
  To demonstrate an improvement from baseline in the parameter left ventricular end-diastolic volume (LVEDV) associated with the Carillon Mitral Contour System (Intervention group) relative to the Control group.
Secondary Efficacy Objective 3 - Change in LV End-Systolic Volume | 12 months
  To demonstrate an improvement from baseline in the parameter left ventricular end-systolic volume (LVESV) associated with the Carillon Mitral Contour System (Intervention group) relative to the Control group.
Secondary Efficacy Objective 4 - Change in 6 Minute Walk Distance | 12 months
  To demonstrate a significantly greater improvement from baseline in six-minute walk distance associated with the Carillon Mitral Contour System (Intervention group) relative to the Control group.
Secondary Efficacy Objective 5 - Change in KCCQ | 12 months
  To demonstrate the improvement from baseline in the overall summary score of the Kansas City Cardiomyopathy Questionnaire (KCCQ) associated with the Carillon Mitral Contour System (Intervention group) relative to the Control group.
Secondary Efficacy Objective 6 - Change in NYHA Classification | 12 months
  To demonstrate the improvement in the proportion of patients who improve by at least one NYHA class from baseline associated with the Carillon Mitral Contour System (Intervention group) relative to the Control group.
Secondary Efficacy Objective 7 - Percent days lost due to HFH or CV death | 12 months of follow-up, and any available data up to 24 months
  To compare percent days lost due to HFH and CV death, relative to Control, analyzed when the last subject completes 12 months of follow-up and use all available data up to 24 months.
Secondary Efficacy Objective 8 - Incidence of alternative therapy and all-cause mortality | 12 months of follow-up, and any available data up to 24 months
  To compare the incidence of need for alternative therapy and all-cause mortality (superiority test if HR < 1), relative to Control, analyzed when the last subject completes 12 months of follow-up and use all available data up to 24 months
Secondary Efficacy Objective 9 - Total number of HFH | 12 months of follow-up, and any available data up to 24 months
  To compare total number of HFH, relative to Control, analyzed when the last subject completes 12 months of follow-up and use all available data up to 24 months
Secondary Safety Objective - Freedom from peri-procedural Major Adverse Events | 30 days or hospital discharge date, whichever is longer
  Freedom from a composite of major adverse events (defined as Death, Myocardial Infarction, Device Embolization, Vessel Erosion, Cardiac Perforation, and occurrence of cardiac surgery or percutaneous coronary intervention) in the Intervention group is greater than 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kapadia, MD, Principal Investigator — The Cleveland Clinic; Randall Starling, MD, Principal Investigator — The Cleveland Clinic
Locations (74):
- United States (62):
  - Dignity Health Research Institute at Mercy Gilbert and Chandler Regional Medical Centers, Gilbert, Arizona
  - Banner Health - Phoenix, Phoenix, Arizona
  - Tucson Medical Center Health, Tucson, Arizona
  - Banner University Tuscon, Tucson, Arizona
  - Memorial Care Hospital, Long Beach, California
  - Keck School of Medicine of USC, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Redwood City, California
  - Scripps Health, San Diego, California
  - University of California- San Francisco, San Francisco, California
  - South Denver Cardiology, Littleton, Colorado
  - Medstar, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - University of Miami, Miami, Florida
  - Advent Health Hospital, Orlando, Florida
  - Palm Beach Gardens Medical, Palm Beach, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Augusta University Research Institute, Augusta, Georgia
  - Wellstar Health System,, Marietta, Georgia
  - Advocate Good Samaritan, Downers Grove, Illinois
  - Midwest Cardiovascular Institute (MCI), Naperville, Illinois
  - Prairie Heart Institute, Springfield, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Cardiovascular Institute South, Houma, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - St Elizabeth's Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. Marys Research Institute, Saginaw, Michigan
  - CentraCare Heart and Vascular, Saint Cloud, Minnesota
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Deborah Heart & Lung, Browns Mills, New Jersey
  - Hackensack University Medical Center, Edison, New Jersey
  - Albany Medical College,, Albany, New York
  - University at Buffalo, Buffalo, New York
  - Vassar Brothers- Hudson Valley Cardiovascular Practice, Poughkeepsie, New York
  - Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - Harrington Vascular, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Kettering Health Research Institute, Dayton, Ohio
  - Oklahoma Heart Institute Hospital, Tulsa, Oklahoma
  - Saint Francis Hospital,, Tulsa, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Providence Heart Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn Medicine Lancaster General Health, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Lankenau Institute of Medical Research, Wynnewood, Pennsylvania
  - North Central Heart-Avera, Sioux Falls, South Dakota
  - Centennial Medical Center, Nashville, Tennessee
  - Houston Healthcare Medical Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Henrico Doctors Hospital, Henrico, Virginia
  - HCA Chippenham Medical Center, Richmond, Virginia
  - Carilion Hospital, Roanoke, Virginia
  - Advocate Aurora Research Institute, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - St Boniface Hospital - University of Manitoba, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
  - Unity Health Toronto, St Michael's Hospital, Toronto, Ontario
- France (5):
  - Pole Sante Republique, Clermont-Ferrand
  - Centre Hospitalier Universitaire De Lille, Lille
  - Hôpital Cardiologique Louis Pradel, Lyon
  - Clinique du Millènaire Montpelier, Montpellier
  - Hôpital Européen Georges-Pompidou, Paris
- European Interbalkan Medical Center, Thessaloniki, Greece
- Poznan University of Medical Sciences, Poznan, Poland
- St James University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schofer J, Siminiak T, Haude M, Herrman JP, Vainer J, Wu JC, Levy WC, Mauri L, Feldman T, Kwong RY, Kaye DM, Duffy SJ, Tubler T, Degen H, Brandt MC, Van Bibber R, Goldberg S, Reuter DG, Hoppe UC. Percutaneous mitral annuloplasty for functional mitral regurgitation: results of the CARILLON Mitral Annuloplasty Device European Union Study. Circulation. 2009 Jul 28;120(4):326-33. doi: 10.1161/CIRCULATIONAHA.109.849885. Epub 2009 Jul 13. PMID 19597051
- [Background] Siminiak T, Wu JC, Haude M, Hoppe UC, Sadowski J, Lipiecki J, Fajadet J, Shah AM, Feldman T, Kaye DM, Goldberg SL, Levy WC, Solomon SD, Reuter DG. Treatment of functional mitral regurgitation by percutaneous annuloplasty: results of the TITAN Trial. Eur J Heart Fail. 2012 Aug;14(8):931-8. doi: 10.1093/eurjhf/hfs076. Epub 2012 May 21. PMID 22613584
- [Background] Lipiecki J, Siminiak T, Sievert H, Muller-Ehmsen J, Degen H, Wu JC, Schandrin C, Kalmucki P, Hofmann I, Reuter D, Goldberg SL, Haude M. Coronary sinus-based percutaneous annuloplasty as treatment for functional mitral regurgitation: the TITAN II trial. Open Heart. 2016 Jul 8;3(2):e000411. doi: 10.1136/openhrt-2016-000411. eCollection 2016. PMID 27493761